CLINICAL TRIAL: NCT00136461
Title: A Randomized Phase II Trial of All-Trans Retinoic Acid and One of Two Schedules of Bryostatin 1 in Patients With Refractory Acute Myelogenous Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Brief Title: A Study of All-Trans Retinoic Acid (ATRA) and Bryostatin in Patients With Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 96-278; NCI# T96-0112
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: AML; acute myelogenous leukemia; MDS; myelodysplastic syndrome; bryostatin 1; all-trans retinoic acid; ATRA
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Tretinoin; bryostatin 1

INTERVENTIONS:
Drug: All-trans retinoic acid
Drug: Bryostatin 1

SUMMARY:
The purpose of this study is to assess the effects of the combination of all-trans retinoic acid in combination with one of two schedules of Bryostatin 1 in patients with myelodysplasia and acute myelogenous leukemia.

DETAILED DESCRIPTION:
All patients receive all-trans retinoic acid at a dose of 150 mg/m2/day and patients are randomized to one of two schedules of Bryostatin 1.

Arm 1: Bryostatin 1 is administered at a dose of 60 mcg/m2 as a 30 minute intravenous (IV) infusion on days 8 and 22.

Arm 2: Bryostatin 1 is administered at a dose of 40 mcg/m2 as a 72 hour IV infusion starting on days 8 and 22.

Patients are assessed for response on day +50 with a bone marrow examination and patients with either a clinical response or stable disease receive further therapy.

Bryostatin 1 pharmacokinetic samples are to be drawn on days 1, 8 and 50 of each cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML who have failed induction chemotherapy.
* Patients with secondary AML
* Patients with AML over age 60 who are deemed not to be a candidate for chemotherapy.
* Patients with any subtype of MDS.
* Age 18 or greater.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Satisfactory liver and kidney function.
* Greater than 4 weeks from prior chemotherapy or radiation therapy.

Exclusion Criteria:

* Central nervous system abnormality.
* Uncontrolled active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 1997-05; Primary Completion 2000-08 (Actual); Study Completion 2000-08 (Actual)

PRIMARY OUTCOMES:
This study is designed to test the therapeutic effect of combining Bryostatin 1 with the known maximum tolerated dose of all-trans retinoic acid in patients with either MDS or AML.

SECONDARY OUTCOMES:
This study will also determine the ability of Bryostatin 1 in combination with ATRA in humans to induce differentiation of human leukemic cells and to cause changes in the levels of protein kinase C isoenzymes in these cells.

CONTACTS AND LOCATIONS:
Overall Officials: Richard M. Stone, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States